CLINICAL TRIAL: NCT05183815
Title: Effectiveness of Slow Back Stroke Massage and Murrotal Quran on Fatigue and
Brief Title: Effectiveness of Slow Back Stroke Massage and Murrotal Quran on Fatigue and Quality of Life of Patients Undergoing Haemodialysis
Acronym: EMQ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Muhammadiyah Yogyakarta (Other)
Responsible Party: Principal Investigator, Erna Rochmawati, Associate Professor, Universitas Muhammadiyah Yogyakarta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMYogyakarta
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Fatigue; Hemodialysis; Chronic Kidney Disease; Quality of Life
MeSH Terms: conditions — Fatigue; Renal Insufficiency, Chronic | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- massage (Experimental)
  Interventions: Other: slow stroke massage and murrotal quran

INTERVENTIONS:
Other: slow stroke massage and murrotal quran — murrotal quran and slow stroke massage
  Other Names: massage

SUMMARY:
The study aimed to investigate the effectiveness of slow back stroke massage and murrotal Quran on fatigue and quality of life on patients undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing hemodialysis minimal 6 months

Exclusion Criteria:

* patients with hear impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-25 (Estimated); Primary Completion 2022-03-10 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Level of Fatigue | 4 weeks
  level of fatigue
Level of quality of life | 4 weeks
  level of quality of life

IPD SHARING:
Plan to Share IPD: Undecided
The researcher will share data based upon request